CLINICAL TRIAL: NCT02706574
Title: Brain Injury Assessment Study at Hennepin County Medical Center
Acronym: BASH
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: CentraCare (Other)
Collaborators: Abbott Diagnostics Division (Industry)
Responsible Party: Sponsor
Other Study IDs: HSR 15-4079
Record Dates: First submitted 2016-02-29; First posted 2016-03-11 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Traumatic Brain Injury
Keywords: Eye Tracking; Blood-based Biomarkers; CSF-based Biomarkers; Magnetic Resonance Imaging; Computed Tomography Scan; Outcome Measures
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood draws will be taken for both proteomic and genetic analysis at acute and follow-up time points. The specimens will be used to test a specific set of biomarkers related to traumatic brain injury, and they will also be retained for future discovery efforts of novel biomarkers.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Isolated Traumatic Brain Injury: This group will present to our Level 1 Trauma Center with a Traumatic Brain Injury and no other associated injuries. They will be older than age 4, have no major neurologic or psychiatric disorder, be developmentally normal, and will not be prisoners.
- Isolated Body Trauma: This group will present to our Level 1 Trauma Center as a trauma patient with no injury to their head. They will be older than age 4, have no major neurologic or psychiatric disorder, be developmentally normal, and will not be prisoners.
- Combined Traumatic Brain Injury and Body Trauma: This group will present to our Level 1 Trauma Center as a trauma patient that had injuries to both their head and body. They will be older than age 4, have no major neurologic or psychiatric disorder, be developmentally normal, and will not be prisoners.
- Healthy, Uninjured Controls: This group will consist of subjects that have not been exposed to any major trauma in the previous 12 months. They will be older than age 4, have no major neurologic or psychiatric disorder, be developmentally normal, and will not be prisoners.

SUMMARY:
The goals of this study are to develop an objective, multi-modal classification scheme and outcome measures for traumatic brain injury based on several measures: (1) blood-based biomarkers (indicates which cell types are damaged), (2) eye tracking (detects mass effect/elevated intracranial pressure and pathway disruption), (3) radiographic measures of CT and MRI (detect structural abnormalities), and (4) standardized outcome assessments.

DETAILED DESCRIPTION:
Background:

Current algorithms for assessment of the severity of brain injury include Glasgow Coma Scale score and other measures. These measures are adequate for relating acute severity but are insufficiently sensitive for subtle pathology which can result in persistent deficit. The Glasgow Coma Scale (GCS) and other measures also do not enable differentiation among types of injury. Thus patients grouped into a single GCS level entering a clinical trial may have vastly heterogeneous severity and type of injury. Because outcomes also vary accordingly, inappropriate classification undermines the integrity of a clinical trial. Improved classification of injury will enable more precise delineation of disease severity and type for patients with a traumatic brain injury (TBI) in clinical trials.

Additionally, current brain injury trials rely on outcome measures such as Glasgow Outcome Scale Extended, which capture global phenomena but fail to assess for subtle differences in outcome. Thus, many recent trials for brain injury therapeutics have failed. Sensitive outcome measures are needed to determine how well patients have recovered from brain injury in order to test therapeutics and prophylactics.

Overview of Methods:

All trauma patients that span the full spectrum ranging from non-brain injured, to CT-negative, to structurally brain injured, requiring surgery will be included in this study. A total of 1000 patients and 200 controls will be recruited over approximately 2 years.

The study has been approved by the Institutional Review Board (IRB), enabling a waiver of consent for all trauma patients until it becomes appropriate to obtain consent. The trauma patients will be screened upon admission, and potentially during the period of waived consent, for participation in the study (target N for screening = 16,000 per year). The screening process will include:

1. A standardized history and physical examination done as a part of the standard of care.
2. A standardized assessment to be done by research personnel.
3. Eye tracking.
4. Analysis of serum biomarkers at three time points within the first 24 hours.
5. MRI scans for a subset of patients within one week of their injury.
6. CT scans as clinically indicated.
7. Pathologic specimen as clinically indicated.
8. Cerebrospinal fluid (CSF) analysis in patients that receive a ventriculostomy catheter.
9. Brain tissue oxygenation analysis in patients receiving Licox.

The screening process that takes place, potentially during the period of waived consent, will allow for patients to be stratified into the following groups with the associated targeted sample sizes over two years:

1. Isolated TBI (N=400)
2. Combined TBI and Body Trauma (N=400)
3. Isolated Body Trauma (N=200)
4. Healthy, Uninjured Controls (N=200)

Upon discharge, patients will be recruited to enroll in a long-term follow-up assessment. They will be seen in the hospital at the following time points post-injury: 2 weeks, 4 weeks, 3 months, 6 months, and 1 year. At these follow-up visits, participants will be asked to undergo various assessments depending on the follow-up visit, including:

1. Eye Tracking.
2. Blood draw for blood-based biomarker analysis.
3. MRI scan if they had one within one week post-injury.
4. CT scan if they had one at admission.
5. Cognitive, Neurologic, and Quality of Life Assessments

Data Analysis:

Patient outcomes, measured with sensitive outcome measures, will be linked to acute research findings in order to create a classification scheme for brain injury that is based on objective measures and can accurately predict prognosis.

ELIGIBILITY:
Inclusion Criteria:

* All trauma patients that present to Hennepin County Medical Center.

Exclusion Criteria:

* Age > 4 years old;
* Major psychiatric or neurologic disorder: Active Psychotic Break, Trauma due to Suicide Attempt, Epilepsy, Multiple Sclerosis, Dementia, Guillain Barre Syndrome/Chronic Inflammatory Demyelinating Polyneuropathy, Significant Neurodegenerative Disorders, Muscular Dystrophy, and/or Malignant Intracranial Mass with Significant Mass Effect.
* Developmentally Abnormal, or
* Prisoners.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will include all trauma patients that present to the HCMC Emergency Department, trauma bay or as a direct transfer to neurosurgery.
Sampling Method: Probability Sample
Enrollment: 774 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Change in Metrics of Eye Movements during Recovery as Measured by Eye Tracking | Post-Injury Time Points of Data Collection: 2 weeks, 4 weeks, 3 months, 6 months, and 1 year.
  Patients will watch a video for 220 seconds as it moves clockwise around the perimeter of a monitor at about 10 seconds per side, resulting in 5 complete rotations of 40 seconds each. As the patient watches the video, their eye movements will be recorded by a camera.
Change in Proteomic Concentrations of Blood-Based Biomarkers during Recovery as Measured by Blood Draws | Post-Injury Time Points of Data Collection: 2 weeks, 4 weeks, 3 months, 6 months, and 1 year.
  Blood will be drawn for proteomic analysis at each follow-up time point. Blood will also be drawn acutely for genomic analysis.
Change in Observable Neural Abnormalities as measured by Magnetic Resonance Imaging | Post-Injury Time Points of Data Collection: within 1 week and at 1 year.
  A group of patients will be selected based on presenting symptoms to undergo a MRI within a week of their injury and again 1 year after their injury. The sequences for these scans will include T2 Flair, susceptibility weighted imaging, diffusion weighted imaging, and diffusion tensor imaging.
Computed Tomography Scan | Post-Injury Time Point of Data Collection: 1 year.
  A group of patients that had an acute CT scan at admission will be selected based on presenting symptoms to undergo a CT scan at 1 year post-injury.

SECONDARY OUTCOMES:
Change in Neurological Examination during Recovery as Measured by the Neurological Outcome Scale after Traumatic Brain Injury | Post-Injury Time Points of Data Collection: 2 weeks, 4 weeks, 3 months, 6 months, and 1 year.
  The Neurological Outcome Scale for Traumatic Brain Injury is a standardized neurological examination validated specifically for patients with Traumatic Brain Injury.
Change in Cognitive Function and Symptom Severity during Recovery as Measured with the Sports Concussion Assessment Tool 3 (SCAT3) | Post-Injury Time Points of Data Collection: 2 weeks, 4 weeks, 3 months, 6 months, and 1 year.
  The Standardized Assessment of Concussion and Symptom Severity Scale subscores of the SCAT3 will be done at every follow-up time point to assess cognitive functioning and symptom severity, respectively, as the patients' recovery progresses.
Change in Quality of Life during Recovery as Measured with the Mayo-Portland Adaptability Inventory-4 (MPAI-4) | Post-Injury Time Points of Data Collection: 3 months, and 1 year.
  The MPAI-4 is a standardized and comprehensive quality of life assessment that will be used to assess self-reported quality of life as the patients' recovery progresses.
Change in Global Outcome during Recovery as Measured with the Glasgow Outcome Scale-Extended (GOS-E) | Post-Injury Time Points of Data Collection: 3 months, 6 months, and 1 year.
  The GOS-E is commonly used in traumatic brain injury research to assess global changes in disability following traumatic brain injury as the patients' recovery progresses.
Change in Memory Performance during Recovery as Measured with the Galveston Orientation and Amnesia Test (GOAT) | Post-Injury Time Points of Data Collection: 3 months and 1 year.
  The GOAT is commonly used in traumatic brain injury research to assess global changes in memory performance following traumatic brain injury as the patients' recovery progresses.
The Number of Prior Brain Injuries the Patient has Suffered as Measured with the Boston Assessment of Traumatic Brain Injury-Lifetime | Post-Injury Time Point of Data Collection: 2 weeks.
  This comprehensive and validated tool will allow for an accurate assessment of how many prior brain injuries a patient has had.
Change in Cognitive Functioning during Recovery as Measured by the Brief Test of Adult Cognition by Telephone | Post-Injury Time Points of Data Collection: 3 months and 1 year.
  This test of cognitive function will be used for those patients that are not able to come to the hospital for follow-up assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Uzma Samadani, MD, PhD, Principal Investigator — Physician, Neurosurgery

REFERENCES:
- [Background] Samadani U. A new tool for monitoring brain function: eye tracking goes beyond assessing attention to measuring central nervous system physiology. Neural Regen Res. 2015 Aug;10(8):1231-3. doi: 10.4103/1673-5374.162752. No abstract available. PMID 26487847
- [Background] Samadani U, Ritlop R, Reyes M, Nehrbass E, Li M, Lamm E, Schneider J, Shimunov D, Sava M, Kolecki R, Burris P, Altomare L, Mehmood T, Smith T, Huang JH, McStay C, Todd SR, Qian M, Kondziolka D, Wall S, Huang P. Eye tracking detects disconjugate eye movements associated with structural traumatic brain injury and concussion. J Neurotrauma. 2015 Apr 15;32(8):548-56. doi: 10.1089/neu.2014.3687. Epub 2015 Feb 6. PMID 25582436
- [Background] Samadani U, Farooq S, Ritlop R, Warren F, Reyes M, Lamm E, Alex A, Nehrbass E, Kolecki R, Jureller M, Schneider J, Chen A, Shi C, Mendhiratta N, Huang JH, Qian M, Kwak R, Mikheev A, Rusinek H, George A, Fergus R, Kondziolka D, Huang PP, Smith RT. Detection of third and sixth cranial nerve palsies with a novel method for eye tracking while watching a short film clip. J Neurosurg. 2015 Mar;122(3):707-20. doi: 10.3171/2014.10.JNS14762. Epub 2014 Dec 12. PMID 25495739